CLINICAL TRIAL: NCT04960332
Title: Effect of Negative Pressure Wound Therapy After Surgical Removal of Deep-Seated High-Malignant Soft Tissue Sarcomas of the Extremities and Trunk Wall. A Randomized Controlled Trial
Brief Title: Effect of Negative Pressure Wound Therapy After Surgical Removal of Deep-Seated High-Malignant Soft Tissue Sarcomas of the Extremities and Trunk Wall.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Andrea Thorn, PhD student and Medical Doctor, department of orthopedic surgery, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prevena-RH-2021
Record Dates: First submitted 2021-05-26; First posted 2021-07-13 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Sarcoma; Cancer; Neoplasms, Connective and Soft Tissue
Keywords: Negative Pressure Wound Therapy; Prevena; Sarcoma; Cancer; Neoplasms, Connective and Soft Tissue
MeSH Terms: conditions — Sarcoma; Neoplasms; Neoplasms, Connective and Soft Tissue

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment (No Intervention): Group A: Standard wound closure with staples and conventional wound dressing.
- Prevena (Experimental): Group B: Wound closure with staples and Negative Pressure Wound Therapy (PREVENA PLUS™ Incision Management System).
  Interventions: Device: Prevena

INTERVENTIONS:
Device: Prevena — RCT (no blinding) where the patients will be randomized to wound closure with staples and either Negative Pressure Wound Therapy (PREVENA PLUS™ Incision Management System) for 7 days or a conventional wound dressing.
  Arms: Prevena

SUMMARY:
The purpose of this research project is to improve the surgical treatment of Soft Tissue Sarcoma (STS) treatment based upon a Randomized Controlled Trial (RCT). We want to evaluate the effect of the use of Negative Pressure Wound Therapy (NPWT) versus a conventional wound dressing on postoperative wound complications after surgical removal of deep-seated high-malignant STS of the extremities or trunk wall.

DETAILED DESCRIPTION:
Introduction

Sarcomas are a heterogeneous group of rare malignant tumors of mesenchymal cell origin in the musculoskeletal system comprising 1% of all adult cancers. The reported incidence of all types of sarcomas is approximately six to eight per 100,000 inhabitants corresponding to 300 cases per year in Denmark (250 STS (100 retroperitoneal/abdominal STS), 50 bone sarcomas). Sarcomas arise in the body's connective tissues including bone, muscle, cartilage, fat tissue, blood vessels, and peripheral nerve-sheaths and hence arise in all parts of the body although most dominant in the extremities (78%).

There exist more than 50 histologic subtypes of STS yielding a broad heterogeneous morphology and biological behavior of all subtypes. The incidence of STS is in general increasing with age (median age=65). High-grade soft tissue sarcomas mostly metastasize hematogenous to the lungs, which is also the primary cause of sarcoma-specific death and approximately 10% of patients with STS have metastases at diagnosis.

Treatment of STS requires a multidisciplinary highly specialized team, evaluating risks and benefits of all available options and expected outcomes with the aim to minimize the recurrence of disease and preserve function and quality of life. The main treatment principles that have largely been unchanged since the 1980ies is surgery supplemented with adjuvant radiotherapy depending on subtype and stage. The use of NPWT after high-risk orthopedic surgeries such as e.g. amputations, treatment of open fractures and joint replacement surgery are increasing, but the direct cost is much higher compared to the conventional wound dressing. However, previous studies have shown that NPWT can reduce postoperative complications such as wound dehiscence and infection. STS surgery that is often combined with pre-or postoperative radiation therapy is a high-risk procedure concerning wound complications and postoperative infections. A retrospective study showed that NPWT reduced the risk of wound complications in patients with lower extremity STS treated with preoperative radiation and the use of NPWT was not associated with an increased risk of local recurrence.

Methods

Study design

RCT (no blinding) where the patients will be randomized to wound closure with staples and either NPWT (PREVENA PLUS™ Incision Management System) for 7 days or a conventional wound dressing.

Randomization

All 160 patients will in the operating room be randomized (randomization with 80 in each group) to receive one of the two treatment:

Group A: Standard wound closure with staples and conventional wound dressing. Group B: Wound closure with staples and NPWT (PREVENA PLUS™ Incision Management System).

Block randomization with 8 patients in each block stratified for upper extremity/truncal wall or lower extremity STS verified using a computerized irreversible application - the Research Electronic Data Capture (REDCap). The randomization sequence will be computer-generated.

Institutions

- Department of Orthopedic Surgery, Rigshospitalet, University of Copenhagen and Department of Orthopedic Surgery, Aarhus University Hospital: The surgeries will be performed in these two department, both are tertiary multidisciplinary center performing highly specialized tumor surgeries.

Materials

Patients

Identification and inclusion Patients evaluated at a multidisciplinary conference and afterward with a biopsy verified STS will be identified in Sundhedsplatformen (electronic patient journal), the only information needed from the patient journal prior informed consent is when they will meet in the outpatient clinic. Patients eligible for inclusion will at their first outpatient visit to plan further final surgery be informed about the study written and orally. On the day of their surgery written informed consent will be obtained if they want to participate in this study. No patient will have below 48 hours to answer, complied with the Helsinki declaration.

All patients will be informed orally and written by the principal investigator, information will be given in a separate room allocated for only the patient and if wanted the assessor, so interruption occurs. All patient will be asked if they want an assessor and so a new meeting will be allocated and the information will again in a separate room allocated for the patient and the assessor be given by the principal investigator.

The written informed consent gives the principal investigator, sponsor and sponsor's representatives as well as any control authority direct access to obtain information in the patient's medical record, etc., including electronic medical record, in order to see information about the subject's health, which is necessary in carrying out the research project and for control purposes, including self-monitoring, quality control and monitoring, which they are required to perform.

The participants are covered by the Danish Patient Compensation Association.

Research plan

1. Clinical wound follow-up (n=160): preoperatively, 7 days, time for removal of staples and 4 months after surgery. To all examinations, clinical photos of the wound will be taken and stored in Sundhedsplatformen (electronic patient journal).
2. Clinical function evaluation (n=160): Musculoskeletal Tumor Society Score (MSTS) and Toronto Extremity Salvage Score (TESS) 4 months and 1 year postoperatively.

Follow-up

Patient's wounds will be followed with photo documentation on day 0, day 7, at definitive wound healing (removal of staples), 4 months postoperatively and in case of major wound complication by a member of the department staff or research group.

Follow-up from day 7 and further on will be performed in the outpatient regime, at Rigshospitalet, orthopedic department or the ortopedic department at Aarhus University Hospital, patients will be convened through e-boks and if necessary, transport will be provided.

Calculation of sample size

In the study of O'Sullivan et al. a major wound complication within 4 months postoperatively was identified in 16 out of 94 (17%) in the group of STS patients treated with surgery and postoperative radiation therapy. There exist no studies evaluating the effect of NPWT on wound complications after surgery for STS combined with postoperative radiation therapy. However, in retrospective studies it was found that NPWT reduced the risk of wound complications from 47% to 8% (83% reduction) in patients with lower extremity STS treated with preoperative radiation [14] and from 27% to 7% (75% reduction) in patients undergoing hip and knee revision surgery.

In a study design with an 80% risk of avoiding type II error, a 5% risk of type I error and an 80% wound complication risk reduction in a population similar to the study by O'Sullivan et al. the investigators will need to include 154 STS patients (77 in each group) in an RCT.

To make allowance for dropouts (since the follow-up period regarding the primary study endpoint is only 4 months = 120 days few dropouts are expected) during the study period the investigators plan to include 160 patients.

Risks, side effects and disadvantages

The investigators do not expect that the patients participating in the study will experience any special side effects or complications related directly to the specific use of NPWT or the standard wound closure. The dressing may for some patients give a mild skin irritation of the skin under the enclosed dressing or a slight discomfort with having to wear an occlusive dressing. Any skin irritation that is transient (i.e., resolves within 24 hours following device use and requires no medical intervention), will not be classified as an adverse device effect. Some blistering formations have been reported in relation to total hip and knee replacement surgery, but no more than tape trauma in patients with conventional dressing.

A retrospective study showed that NPWT reduced the risk of wound complications in patients with lower extremity STS treated with preoperative radiation and the use of NPWT was not associated with an increased risk of local recurrence.

No risk or side effects are reported by the manufacture when adhering to the manual of use.

Prevena™ NPWT are used daily at the orthopedic department, it is a CE classified medical devised and due to use in the recommended field approval from danish medicines agency are not necessary.

Ethical considerations

Approval from the Scientific Ethical Committee (H-21013549) and the Data Protection Agency (P-2021-150) has been obtained and the study is registered at clinicaltrial.gov NCT04960332. All patients will receive both oral and written information before written informed consent to participate is obtained.

The regulation from data protection regulation and data protection act will always be followed and a permission from data protection agency have been obtained (P-2021-150).

The significant use of the present study is new knowledge concerning the best way to treat a certain group of patients with deep-seated STS of an extremity or the trunk wall. Knowledge from our study will benefit society in general, and optimize utilization of resources, in terms of the best treatment for future patients.

In case of serious adverse preliminary results, data will be analyzed and if one of the treatments is found to cause significant critical problems compared to the other (p<0.05), the study will be ended. The study is thus designed to minimize unnecessary risks to the patients.

Statistical analysis

Fisher's exact test will be used for categorical variables. Depending on if the data could be considered normally distributed or not, a t-test for unpaired data or Mann-Whitney U test will be used for continuous variables.

Kaplan Meier survival analysis for overall survival (with log-rank test for comparison of groups). In case of an assumption of a difference in time to delayed wound healing, competing risk analysis will be used to address differences between the groups with death and amputation as competing factors.

All analyses will be performed in accordance with the intention-to-treat principles.

Two-sided p-values below 0.05 will be considered statistically significant.

Time frame

According to the latest report from the Danish Sarcoma Registry, there were approximately 900 newly diagnosed sarcomas in Eastern Denmark (Rigshospitalet) during the 5 years from 2014 to 2018. The majority, but not all of the patients are suffering from high-malignant deep-seated STS of the extremities or the trunk wall. The inclusion of patients in the study will start at the first half of of 2021 thus leaving at least 3 years for inclusion and reserve 6 months for the PhD-student to do data management and writing.

ELIGIBILITY:
Inclusion Criteria:

- Surgery for a deep-seated STS of an extremity or the trunk wall at Rigshospitalet.

Exclusion Criteria:

* Age < 18 years
* Wound closure not possible without plastic surgery (pedicled or free flaps)
* Low malignant (Trojani grade 1) STS or borderline tumors
* Pre- or postoperative chemotherapy
* Preoperative radiotherapy to the local site.
* Allergic or hypersensitive to acrylic adhesives or silver
* Unwilling or unable to provide informed consent
* Inability to comply with planned study procedures
* Patients with metastatic disease.
* Patients with ischemic surgery such as bypass or endovascular prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Wound complication/healing | 120 days postoperatively
  A major wound complication defined as in O'Sullivan et al. [11]:
  * A secondary surgery under anesthesia for wound repairs such as debridement, operative drainage and secondary wound closure.
  * Wound management without secondary surgery, this includes invasive procedure without anesthesia such as aspiration of seroma and readmission for wound care such as intravenous antibiotic or persistent deep packing within 4 months (120 days) after surgery.

SECONDARY OUTCOMES:
Secondary outcome measures, hospital stay. | 1 year postoperatively
  Length of hospital stay (measured in days)
Secondary outcome measures, readmission. | 1 year postoperatively
  Readmission to hospital for treatment of a wound complication (measured in days from primary surgery)
Secondary outcome measures, primary wound healing. | 1 year postoperatively
  Time to primary wound healing and removal of staples, ready for radiation therapy (measured in days from primary surgery)
Secondary outcome measures, deep infection. | 1 year postoperatively
  Deep infection (measured in days from primary surgery, any medical or surgical interventions will be described)
Secondary outcome measures, seroma. | 1 year postoperatively
  Postoperative seroma development (measured in days from primary surgery)
Secondary outcome measures, MSTS. | 1 year postoperatively
  Musculoskeletal Tumor Society Score (MSTS)
  MSTS score is a physician-completed score containing following categories:
  * Pain
  * Function
  * Emotional acceptance
  * Support/Assistive device
  * Walking
  * Gait
  Maximum score is 30 (the value will often be presented in percentage of total).
Secondary outcome measures, TESS. | 1 year postoperatively
  Toronto Extremity Salvage Score (TESS)
  TESS is a self-administrated questionnaire that evaluates physical disability, it consists of 29 questions for upper-extremity and 30 for lower-extremity. Each question is scored from 1-5, where 5 is given if there are no problems. Values will often be presented as a percentage of the total possible amount.
Secondary outcome measures, 5Q-5D. | 1 year postoperatively
  European Quality of Life - 5 Dimensions (EQ-5D)
  EQ-5D is a self-reported questionnaire to evaluate the quality of life, it has 5 dimensions:
  * Mobility
  * Personal hygiene
  * Usual activities
  * Pain
  * Anxiety/depression Each dimension is evaluated with a score of 1-5, where 1 is given to patients without problems. Each answer has a different weight in values and the values for a Danish population will be used in analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Thorn, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No
The regulation from data protection regulation and data protection act will always be followed and a permission from data protection agency have been obtained (P-2021-150).

REFERENCES:
- [Derived] Yilmaz M, Thorn A, Sorensen MS, Jensen CL, Petersen MM. Effect of negative pressure wound therapy after surgical removal of deep-seated high-malignant soft tissue sarcomas of the extremities and trunk wall-study protocol for a randomized controlled trial. Trials. 2022 Jun 18;23(1):507. doi: 10.1186/s13063-022-06468-6. PMID 35717239